CLINICAL TRIAL: NCT00444717
Title: Multicenter Study for Anti-oxidative and Anti-inflammatory Effects of Pitavastatin in Hypercholesterolemic Patients With Metabolic Syndrome
Brief Title: Impact of Pitavastatin in Hypercholesterolemic Patients With Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aichi Gakuin University (Other)
Responsible Party: Tatsuaki Matsubara, Department of Internal Medicine, School of Dentistry, Aichi Gakuin University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGU-64
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2008-10

CONDITIONS: Metabolic Syndrome; Oxidative Stress; Inflammation
Keywords: statin; metabolic syndrome; oxidative stress; inflammation
MeSH Terms: conditions — Metabolic Syndrome; Inflammation | interventions — pitavastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: pitavastatin — Pitavastatin (2mg/day) was administered for 12 weeks
  Other Names: livalo

SUMMARY:
The purpose of this study is to evaluate anti-oxidative and anti-inflammatory effects of pitavastatin in hypercholesterolemic patients with the metabolic syndrome.

DETAILED DESCRIPTION:
The metabolic syndrome is defined as a cluster of cardiovascular risk factors including visceral obesity, dyslipidemia, elevated blood pressure and impaired glucose tolerance. Recently, it has been described that oxidative stress and inflammatory reaction, which are important in progression of atherosclerosis, increases in individuals with the metabolic syndrome. Statins might have beneficial effects such as anti-oxidative and anti-inflammatory actions that are independent from their cholesterol-lowering effects. Pitavastatin, a chemically synthesized statin, has potent LDL-cholesterol lowering and also anti-oxidative and anti-inflammatory effects in animal studies. However, the effects of pitavastatin on oxidative stress and inflammatory action in patients with the metabolic syndrome have not been reported.

ELIGIBILITY:
Inclusion Criteria:

* Hypercholesterolemic patients

Exclusion Criteria:

* Patients receiving lipid-lowering agents
* Familial hypercholesterolemia
* Renal disease
* Diseases of liver, gallbladder and bile ducts
* Pregnant women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Thiobarbituric acid reactive substance; high sensitive C-reactive protein | 12 weeks

SECONDARY OUTCOMES:
Total cholesterol; LDL-cholesterol; HDL-cholesterol; triglyceride; | 12 weeks
Homeostasis model assessment for insulin resistance; adiponectin; | 12 weeks
Soluble intercellular adhesion molecule-1 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuaki Matsubara, MD, PhD, Principal Investigator — Department of Internal Medicine, School of Dentistry, Aichi Gakuin University
Locations (1):
- Tatsuaki Matsubara, Nagoya, Aichi-ken, Japan

REFERENCES:
- [Derived] Matsubara T, Naruse K, Arakawa T, Nakao M, Yokoi K, Oguri M, Marui N, Amano T, Ichimiya S, Ohashi T, Imai K, Sakai S, Sugiyama S, Ishii H, Murohara T. Impact of pitavastatin on high-sensitivity C-reactive protein and adiponectin in hypercholesterolemic patients with the metabolic syndrome: the PREMIUM Study. J Cardiol. 2012 Nov;60(5):389-94. doi: 10.1016/j.jjcc.2012.07.012. Epub 2012 Aug 11. PMID 22884685